CLINICAL TRIAL: NCT05306093
Title: Chronic Effect of a Standardized Saffron Extract on Depressed Mood and Anhedonia in Healthy Adults. A Randomized Controlled Double-blind Clinical Trial.
Brief Title: Depressed Mood and Anhedonia in Healthy Adults
Acronym: MOOD5
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur de Lille (Other)
Responsible Party: Principal Investigator, Jean-Michel Lecerf, Principal investigator, Institut Pasteur de Lille
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2021-A02123-38
Record Dates: First submitted 2022-02-15; First posted 2022-03-31 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Anhedonia; Depressed Mood
Keywords: saffron extract
MeSH Terms: conditions — Anhedonia; Consciousness Disorders | interventions — Dietary Supplements; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutraceutical (Experimental): Daily, 2 dietary supplements will be taken orally with some water, the first one during the breakfast and the second one during the dinner.
  Dietary supplements in capsule form
  Interventions: Dietary Supplement: Nutraceutical
- Maltodextrin (Placebo Comparator): Daily, 2 dietary supplements will be taken orally with some water, the first one during the breakfast and the second one during the dinner.
  Dietary supplements in capsule form
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Nutraceutical — Food supplements are consumed during 8 weeks by healthy volunteers
  Arms: Nutraceutical
Dietary Supplement: Maltodextrin — Food supplements are consumed during 8 weeks by healthy volunteers
  Arms: Maltodextrin

SUMMARY:
The aim of this study is to evaluate the effect of nutraceutical supplement on depressed mood and anhedonia in volunteers after 8 weeks of consumption.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 20 and 65 years (limits included);
* Body Mass Index (BMI) ≥19 and < 30 kg/m²;
* Considered healthy based on their medical history and clinical examination;
* Subjects self-reporting anhedonia based on SHAPS questionnaire. Score ≥ 3 allows the inclusion;
* Subjects with depressive mood disturbance based on POMS depression subscale. Score ≥ 4 allows the inclusion;
* Able and willing to participate to the study by complying with the protocol procedures as evidenced by his dated and signed informed consent form;
* Affiliated with a social security scheme;
* Agreeing to be registered on the national file of the volunteers in biomedical research.

Exclusion Criteria:

* Suffer from mental health other than mild depressive or anxiety symptoms as measured by the Patient Health Questionnaire (PHQ-9). Volunteers with PHQ-9 score >14 could not be included;
* Having suicidal thoughts: score ≥1 at the item 9 of the PHQ-9;
* Diagnosis of medical or psychiatric conditions including (but not limited to):

  * psychiatric disorder (other than mild-to-moderate depression symptoms, anhedonia or anxiety),
  * neurological disease (Parkinson's, Alzheimer's disease, intracranial haemorrhage, head or brain injury),
  * cancer/malignancy,
  * cardiovascular disease (other than hypertension),
  * Immunological disease,
  * endocrine disease (including diabetes or thyroid diseases, Chronic kidney disease, hematological abnormalities);
* Smokers (more than 5 cigarettes per day);
* Uncontrolled hypertension with medication (SBP ≥ 160mmHg or DBP ≥ 100 mmHg) or without medication (SBP ≥ 140mmHg or DBP ≥ 90 mmHg);
* Taking drugs (anxiolytics, antidepressants, antihistamine drug more than 7 day/month) known to have an impact on mental health in the month preceding inclusion and / or likely to consume them during the study and/or Illicit drug;
* Undergoing a psychotherapy in the month preceding inclusion or during the study;
* Consuming more than 3 standard drinks of alcoholic beverage daily;
* Weight change above 10% body weight within the past 6 months before inclusion;
* Currently under prescribed diet regimen, whatever the reason;
* Consuming foods supplement known to have an influence on mental health in the month preceding the inclusion and / or likely to take during the study;
* Consuming more than 50g of chocolate/day;
* For females: Pregnant or planning pregnancy during the study or breastfeeding;
* Any intolerance or allergy documented or suspected to one of the components of the study products;
* Taking part in another clinical trial or being in the exclusion period of a previous clinical trial;
* Subject who would receive more than 4500 euros as indemnities for his participation in biomedical research within the 12 last months, including the indemnities for the present study;
* Under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision;
* Presenting a psychological or linguistic incapability to sign the informed consent and to answer the study questionnaires
* Any other condition which in the investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Mood disturbance evaluated by the Profile Of Mood States (POMS) total score | Baseline (V1)
  The POMS is a self-reported validated questionnaire assessing six mood subscales: tension-anxiety, depression, anger-hostility, vigor, fatigue, and confusion. In our study, a score on POMS depression subscale < 4 does not allow the inclusion.
Mood disturbance evaluated by the Profile Of Mood States (POMS) total score | at 2 weeks
  The POMS is a self-reported validated questionnaire assessing six mood subscales: tension-anxiety, depression, anger-hostility, vigor, fatigue, and confusion. In our study, a score on POMS depression subscale < 4 does not allow the inclusion.
Mood disturbance evaluated by the Profile Of Mood States (POMS) total score | at 4 weeks (V2)
  The POMS is a self-reported validated questionnaire assessing six mood subscales: tension-anxiety, depression, anger-hostility, vigor, fatigue, and confusion. In our study, a score on POMS depression subscale < 4 does not allow the inclusion.
Mood disturbance evaluated by the Profile Of Mood States (POMS) total score | at 6 weeks
  The POMS is a self-reported validated questionnaire assessing six mood subscales: tension-anxiety, depression, anger-hostility, vigor, fatigue, and confusion. In our study, a score on POMS depression subscale < 4 does not allow the inclusion.
Mood disturbance evaluated by the Profile Of Mood States (POMS) total score | at 8 weeks (V3)
  The POMS is a self-reported validated questionnaire assessing six mood subscales: tension-anxiety, depression, anger-hostility, vigor, fatigue, and confusion. In our study, a score on POMS depression subscale < 4 does not allow the inclusion.

SECONDARY OUTCOMES:
Tension, anger, vigour, fatigue and confusion evaluated by the five POMS sub-scores | Baseline (V1) and 1st month (4 weeks (V2)) and between baseline and the end of the study (8 weeks (V3))
  The POMS is a self-reported validated questionnaire assessing six mood subscales: tension-anxiety, depression, anger-hostility, vigor, fatigue, and confusion.
Depression level evaluated by the Center of Epidemiologic Studies Depression scale (CES-D) score | Baseline (V1) and each evaluation (at 1 week, 2 weeks, 3 weeks, 4 weeks (V2), 5 weeks, 6 weeks, 7 weeks and the end of the study : 8 weeks (V3))
  This validated self-reported questionnaire measures levels of depressive symptomatology, with special emphasis on the affective components and depressed mood.
Stress, spleep, anxiety, sadness, energy feeling, attention to others and desire to do things evaluated by Visual Analogic Scales (VAS) score | Baseline (V1) and each week evaluation (1 week, 2 weeks, 3 weeks, 4 weeks (V2), 5 weeks, 6 weeks, 7 weeks and the end of the study : 8 weeks (V3))
  The visual analog scales will be completed by the subjects at V1 and 2 times a week until 8 weeks. Eight dimensions are observed : stress, spleep, anxiety, happiness, energy feeling, irritability, motivation and pleasure.
  Score 0 to 10.
Pleasure feeling evaluated by the Snaith-Hamilton Pleasure Scale (SHAPS) score | Baseline (V1) and each evaluation (2 weeks, 4 weeks (V2), 6 weeks and 8 weeks (V3)
  The Snaith-Hamilton Pleasure Scale (SHAPS) score is a 14-item self-reported validated questionnaire evaluating the pleasure. It covers four domains of hedonic experience: interest/pastimes, social interaction, sensory experience and food/drink.
  A total score can be calculated by adding the responses to each question, ranging from 0 (no anhedonia) to 14 (complete anhedonia).
Quality of life evaluated by the Multicultural Quality of Life Index (MQLI) | Baseline (V1) and 1st month (4 weeks (V2)) and between baseline and the end of the study (8 weeks (V3))
  This validated self-reported questionnaire is composed of 10 items which cover key aspects of the quality of life, from physical well-being to spiritual fulfilment.

CONTACTS AND LOCATIONS:
Overall Officials: Zakaria NAFLI, MD, Principal Investigator — CEN Experimental
Locations (1):
- CEN Experimental, Dijon, France

IPD SHARING:
Plan to Share IPD: No